CLINICAL TRIAL: NCT00315848
Title: A Multi-Center, Randomized, Double-Blind, Parallel Group Study of the Safety and Efficacy of Buprenorphine Transdermal Delivery System Vs. Oxycodone/Acetaminophen Tablets Vs. Placebo in Patients With Chronic Pain Due to Osteoarthritis
Brief Title: The Safety and Efficacy of the Buprenorphine Transdermal Delivery System in Subjects With Osteoarthritis Pain.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Purdue Pharma LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP96-0101
Record Dates: First submitted 2006-04-18; First posted 2006-04-19 (Estimated); Last update posted 2006-05-03 (Estimated); Status verified 2006-04

CONDITIONS: Osteoarthritis
Keywords: chronic pain; osteoarthritis; opioid; transdermal
MeSH Terms: conditions — Osteoarthritis; Chronic Pain

INTERVENTIONS:
Drug: Buprenorphine transdermal delivery system

SUMMARY:
The objective of this study is to demonstrate the effectiveness and tolerability of the buprenorphine transdermal system (5, 10, and 20 mg) in comparison to placebo transdermal system and immediate release oxycodone/acetaminophen in subjects with osteoarthritis pain inadequately treated with non-opioid analgesics. The double-blind treatment intervention duration is 60 days.

DETAILED DESCRIPTION:
Buprenorphine is a synthetic opioid analgesic with over twenty-five years of international clinical experience indicating it to be safe and effective in a variety of therapeutic situations for the relief of moderate to severe pain. Transdermal systems may offer advantages over currently indicated oral products including ease and convenience of use, improved compliance, possible reduction in patient care, and prolonged and consistent delivery of drug.

ELIGIBILITY:
Inclusion Criteria:

* unacceptable pain control despite currently taking a nonsteroidal anti-inflammatory drug considered at a therapeutic and/or tolerated dose or currently taking </=2 short-acting opioid doses per day.
* taking >/=3 opioid doses per day with or without acceptable pain control.

Exclusion Criteria:

* receiving opioids at an average daily dose of greater than 60 mg of oral morphine equivalents or subjects receiving more than 6 tablets per day of a short-acting opioid.
* scheduled to have surgery (including dental) involving the use of post- or preoperative analgesics or anesthetics during the study period.

Other protocol-specific exclusion/inclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225
Dates: Start 1996-11; Study Completion 1999-12

PRIMARY OUTCOMES:
Pain on average and pain right now scores at days 0, 9, 15, 30, 45, 60, or at early termination.

SECONDARY OUTCOMES:
Brief Pain Inventory
dropouts due to lack of efficacy
MOS health survey
VAS pain intensity
therapeutic response
patient preference
daily patient diary
and number of oxycodone/acetaminophen or placebo tablets taken

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Rheumatology Associates of North Alabama, Huntsville, Alabama
  - Arizona Research and Education, Phoenix, Arizona
  - Phoenix Center for Clinical Research, Phoenix, Arizona
  - Western Integrated Pain Treatment Centers, Westminster, Colorado
  - Gainesville Clinical Research Center, Gainesville, Florida
  - Park Place Therapeutic Center, Plantation, Florida
  - MediSphere Medical Research Center, L.L.C., Evansville, Indiana
  - Stratton VA Medical Center, Albany, New York
  - Metroplex Clinical Research Center, Dallas, Texas
  - Arthritis Diagnostic and Treatment Center, San Antonio, Texas